CLINICAL TRIAL: NCT03278236
Title: Does Time Restricted Feeding Improve Glycaemic Control in Overweight Men?
Acronym: RESHAPE2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding to complete pilot.
Sponsor: University of Adelaide (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, A/Prof, University of Adelaide
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HREC/17/RAH/307
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Type2 Diabetes; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRF (Experimental)
  Interventions: Behavioral: TRF

INTERVENTIONS:
Behavioral: TRF — Participants will be instructed to consume their habitual diet within a self-selected 10 hour period every day.

SUMMARY:
Obesity is a serious medical condition, the adverse consequences of which include increased risk of cardiovascular disease, diabetes mellitus, reduced fertility and cancer. The economic cost of obesity was placed at $58 billion dollars in Australia in 2008 [1]. Studies in mice and non-human primates have shown that moderate caloric restriction (CR) increases lifespan and reduces the incidence of cardiovascular disease, cancer, and type 2 diabetes [2]. Reduced risk of chronic diseases is also observed in humans following CR [3]. However, daily CR is difficult to maintain long term, since the body defends against weight loss by inducing "metabolic adaptation"[3] and altering the hormonal appetite response [4]. An emerging number of studies are examining the effects of limiting food intake to prescribed time periods per day, or every other day. Time restricted feeding (TRF) describes a dieting approach where food is available ad libitum, however only for a limited period of time (i.e. 3-12 hours).

This pilot study will examine the effects of restricting daily food intake to within a 10 hour period on glycaemic control, body weight and biomarkers of metabolic health for 6-weeks. This study will build on the existing knowledge base in humans as to whether meal timing, rather than caloric restriction per se, is important to provide the stimulus required to improve metabolic health and reduce risk of chronic disease.

DETAILED DESCRIPTION:
The timing of meals distributed across the wake cycle may play a role in body weight regulation and metabolic health. In rodents, providing an 12 h feeding opportunity during the active phase abrogated the metabolic consequences of a high fat diet, including maintaining leaner body weight and normal glucose homeostasis [5]. In diet-induced obese rodents, switching to a TRF protocol normalised the metabolic milieu by reducing hyperinsulinemia, hepatic steatosis, and inflammation [6]. Interestingly, when lean animals were switched to a TRF high fat diet protocol, which allowed ad libitum access to the high fat diet for 2 consecutive days per week, simulating a "weekend", lean body weights and metabolic profiles were maintained [6]. These studies suggest that following a TRF protocol is of significant benefit to prevent weight gain, and or to normalise the metabolic milieu.

Observational studies of individuals who undertook the Islamic ritual of fasting during the month of Ramadan [7, 8]. Under these conditions, not only is the timing of food intake restricted, but feeding times are switched to non-daylight hours. The outcomes from these observational studies are mixed, but many have observed reduced cardiovascular risk factors [7, 8]. However, beneficial changes in glycaemic profile are more controversial. One study, using continuous glucose monitors, reported there was a change in the pattern of the glycaemic profile, but no change in overall glycaemia [9]. Other studies have noted that fasting glucose levels are increased following Ramadan [7]. Epidemiological evidence shows that individuals who report consuming more of their daily energy intake at the evening meal were more overweight, than those who reported consumed more of their energy intake before lunch[10]. Similarly, eating lunch late in the day (after 15:00 hrs) was predictive of poorer weight loss during a 20-week dietary intervention study [11] and individuals randomized to consume more calories at breakfast had greater weight loss versus those randomized to eat more calories at dinner after 12 weeks [12]. Taken together these data suggest that consuming more calories in the morning may be beneficial for weight management.

Only a limited number of controlled studies have interrogated the effects of TRF in humans [13-15]. The first was a randomised controlled cross-over intervention, where lean individuals were instructed either to consume all of their calories required for weight maintenance over a 4 hour period from 1700-2100h, or as 3 meals/d for 8 weeks. Consumption of the evening meal was supervised within the laboratory, to ensure subjects consumed the entire meal. Significant reductions in body weight and body fat mass, by 1.4 and 2.1 kg respectively, were noted when following the TRF protocol [13]. Despite this small amount of weight loss, fasting blood glucose levels were increased, and TRF resulted in poorer glucose tolerance in response to an oral glucose tolerance test (OGTT) [14]. Thus, consuming a single, large "dinner" meal was detrimental for metabolic health, although no differences in insulin response were noted [14]. Gill et al also examined the effects of 10-11h TRF in 8 men who were overweight and reported an habitual eating pattern that usually spanned at least 14 hours. A 3% body weight loss was observed after 2 months of TRF, and this was maintained for 12 months[16]. It is unclear whether responses may have differed if the food allowance was prescribed at breakfast or lunch times. Finally, healthy, lean male subjects were allowed to eat ad libitum for 13h per day (6am-7pm) for 2 weeks. Participants reported eating significantly less on the TRF versus the control condition, and lost -0.4kg compared with a gain of +0.6kg in the control condition [15]. Whilst this is a minor change in body weight, this pattern is not that atypical of modern eating patterns, and further restriction of eating times, and assessment of obese individuals under these conditions is warranted. The metabolic health impacts were not reported in either of these studies.

Screening visit (S) - (Informed consent, screening questionnaire): Participants will be assessed by a screening questionnaire (provided for review) for risk of type 2 diabetes, and for their diet, medical and exercise history to determine their eligibility. Potentially eligible participants will be invited to attend SAHMRI and have the research protocol explained to them in detail. Informed consent to participate in the study, including a verbal indication that they understand the general study protocol and requirements is then obtained. Routine clinical checks are then performed (weight, height, waist circumference, blood pressure). If participants meet the eligibility criteria, they will be invited to take part in the study.

Baseline assessment and food intake monitoring: In this study, we will use a smartphone-based monitoring and feedback tool (MyCircadianClock app) to monitor the daily pattern of ingestive behaviour, activity and sleep patterns for 1-week, at baseline as well as during weeks 1,3 and 5. This app was developed by our collaborators at Salk Institute, Professor Satchidananda Panda and Dr Emily Manoogian. Participants in our study will be asked to sign up to the MyCircadianClock smartphone app and using the app are asked to take a photograph of any food and drink that they consume, which time stamps when and what was eaten, for later analysis. This app is part of a study conducted by Professor Panda. The Panda lab will share the identifiable data collected through the app from participants of this study, once they have received verification of informed consent from the participant in our study to do so. This is outlined on page 4 of the SIS and consent asked on page 7 of the SIS/consent form. We have attached IRB approval of the MyCircadianClock study, which explains the app in detail.

TRF: Participants will be instructed to consume their habitual diet within a self-selected 10 hour period every day. Outside of the selected eating period, participants are allowed to consume water (encouraged to drink 6-8 glasses per day) and calorie free foods (e.g. sugar-free drinks and chewing gum) as well as black coffee and/or tea. Participants will track their energy intake using the application described above. This will track compliance, and allow us to assess changes in intake.

Metabolic Testing (W0, W6): Participants will be provided with a standardised meal that provides ~30% of their estimated total daily energy requirement (McCains Lasagne, fruit salad, muesli bar) to consume the evening prior to the study visit, by 1930h. They will arrive at 0730 at the Research Unit following a 12 hour overnight fast. Weight, waist and hip circumference and blood pressure will be measured and a 20G cannula inserted into an antecubital vein. A fasting blood sample (20 mL) is drawn for baseline measurements and to assess HbA1c. A second fasting blood sample (20ml) will be taken immediately prior to consuming a standardised 700kcal liquid meal (EnsurePlus ®; 57% CHO, 28 % fat, 15 % protein) (t=0). 6*10 mL blood samples are drawn at 15,30,60,90,120,180 minutes to measure glucose, free fatty acids, insulin, c-peptide and appetite hormones. A total volume of 100 mL blood will be collected at visit 0 and 6; with a total volume of 200 mL collected over 6 weeks. Appetite responses during the meal will be monitored using standardised visual analog scales.

ELIGIBILITY:
Inclusion Criteria:

overweight (BMI >25.0 kg/m2) Waist circumference >102 cm

Exclusion Criteria:

* Personal history of cardiovascular disease, diabetes, major psychiatric disorders, insomnia
* use of prescribed or non-prescribed medications which may affect energy metabolism, gastrointestinal function, weight or appetite (e.g. domperidone and cisapride, anticholinergic drugs (e.g. atropine), androgenic medications (e.g. testosterone), metoclopramide, orlistat, diuretics)
* use of prescribed glucose-lowering/antidiabetic medication (e.g. metformin, DPP4 inhibitors)
* recent weight change in past 3 months, and/or does not habitually eat breakfast
* uncontrolled asthma, current fever, upper respiratory infections
* individuals who regularly perform high intensity exercise (>2 week)
* current intake of > 140g alcohol/week
* current smokers of cigarettes/cigars/marijuana
* current intake of any illicit substance
* current shift worker
* has donated blood within past 3-months
* unable to comprehend study protocol
* does not own a smartphone

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change in glycaemia | 3 hours
  Change in fasting and postprandial blood glucose following a standard meal test

SECONDARY OUTCOMES:
Change in HbA1c | 6 weeks
Change in body weight | 6 weeks
  changes in body weight (kg)
Change in waist and hip circumference | 6 weeks
  changes in waist and hip circumference (cm) and waist:hip ratio
Change in insulin | 3 hours
  changes in fasting insulin and insulin response to a standard meal
Change in gut peptides | 3 hours
  changes in fasting gut peptides and gut peptide responses to a standard meal
Change in cardiovascular risk | 6 weeks
  changes in blood pressure, blood lipids after 6 weeks of intervention
Change in appetite | 3 hours
  changes in measures of appetite in response to a standard meal
Change in food intake | 6 weeks
  Change in quantity and nutritional composition of food intake

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Heilbronn, PhD, Principal Investigator — University of Adelaide
Locations (1):
- Adelaide Medical School, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Food intake data obtained from the MyCircadianApp will be shared between the researchers and the collaborators.
Supporting Information: ICF